CLINICAL TRIAL: NCT03740009
Title: Effects of a Tissue Selective Estrogen Complex (TESC) on Depression and the Neural Reward System in the Perimenopause
Brief Title: Effects of a Tissue Selective Estrogen Complex (TSEC) on Depression and the Neural Reward System in the Perimenopause"
Acronym: Duavee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-2129
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-03

CONDITIONS: Perimenopausal Disorder; Depression
Keywords: Hormone Replacement Therapy; Estrogen; Depression; Mood Disorders; Estrogen Replacement Therapy; Depressive Disorder; Mental Disorders; Hormones; Physiological effects of drugs; Reproductive Control Agents; Tissue Selective Estrogen Complex
MeSH Terms: conditions — Depression; Mood Disorders; Depressive Disorder; Mental Disorders | interventions — bazedoxifene; Estrogens, Conjugated (USP)

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Perimenopausal women, depressed (Experimental): Participants will take Bazedoxifene/Conjugated Estrogen orally for 3 weeks
  Interventions: Drug: Bazedoxifene/Conjugated Estrogen

INTERVENTIONS:
Drug: Bazedoxifene/Conjugated Estrogen — 20 mg bazedoxifene/0.45mg conjugated estrogens tablets
  Other Names: Duavee

SUMMARY:
Using neuroimaging, the investigator will study the effects of estrogen on mood and brain function in perimenopausal women with depression.

DETAILED DESCRIPTION:
Despite decades of clinical research, depression continues to affect 20.9 million Americans each year and remains the leading cause of disability worldwide. Women are twice as likely as men to experience depression, and depression symptoms are particularly common during periods of hormone change. Depression risk increases 14-fold in the two years surrounding menopause, suggesting that hormone changes may cause depression during this time. Past research has shown that estrogen, in particular, plays an important role in depression during the transition to menopause ("the perimenopause") for the following reasons: 1) depression begins when estrogen levels plummet, 2) estrogen therapy reduces depression symptoms, and 3) when perimenopausal women who were treated with estrogen are taken off of estrogen (without their knowledge), their depression returns. Despite clear evidence that estrogen plays a role in depression during the perimenopause (DPM), the investigators don't know how estrogen affects the brain, which is important for developing effective medications to treat DPM and also for determining which patients are most likely to benefit from medication that replaces the estrogen lost during menopause (estrogen replacement therapy).

The investigator received a grant from the National Institutes of Health, which received preliminary support from the Foundation of Hope, to characterize the effect of estrogen replacement therapy on the brain in women with DPM and women without depression ("controls"). The brain pathway affected most by depression is the neural reward circuit, which consists of a number of different brain regions that act in concert to determine a person's response to rewards. Activity in the neural reward circuit depends on estrogen levels and is reduced in people with depression. The investigator's NIH-funded study will be the first to examine how the neural reward circuit is affected by DPM and estrogen replacement therapy. While estrogen replacement therapy acts as an antidepressant, many women elect not to take estrogen and many physicians discourage its use because of the risk of long-term negative health effects, including breast and uterine cancer. A new FDA-approved compound, Duavee, combines estrogen with another medication, bazedoxifene, which protects against breast and uterine cancer while reducing hot flashes. Duavee may therefore be more acceptable to women with DPM and their doctors than estrogen replacement therapy. However, the effects of Duavee on depression and the neural reward circuit have never been tested, and one can't infer that estrogen will have the same antidepressant effects in the presence of bazedoxifene (which partially blocks the effects of estrogen in certain tissues).

The purpose of the proposed project is to 1) test the antidepressant effects of Duavee, and 2) quantify the effects of Duavee on the neural reward circuit. The investigators expect that Duavee will reduce symptoms of depression and increase activity in the neural reward circuit. In this study, the investigators will recruit medically healthy, unmedicated women with DPM and administer Duavee for 3 weeks (a duration that has been shown in previous studies of estrogen replacement to be sufficient for treating depression). Eligibility will be assessed by an initial telephone screen and confirmed by a gynecologic exam, laboratory testing, and an interview about their current and past depression symptoms. Only women with depression that began during the menopause transition (i.e., when they started skipping periods) will be enrolled. Both before and after treatment, women will have a fMRI brain scan to determine the effects of the medication on the neural reward circuit. During the 3-week treatment, women will come into the clinic to have their blood drawn, refill their medication, and answer questions about their mood and menopause symptoms.This study is important because untreated DPM contributes to cardiac deaths. Many women are afraid to use estrogen replacement therapy because of the long-term risk of cancer and yet refuse to take antidepressants for fear of side effects and stigma. Because Duavee addresses the main potential problems of estrogen replacement therapy, this research stands to revolutionize treatment for DPM. The use of estrogen replacement therapy to treat DPM is a relatively new area of research and one of great importance given the large and increasing number of women who enter the perimenopause each year and are potentially at risk for depression. Women with DPM seek treatment from gynecologists, psychiatrists, and general practitioners, yet there is neither consensus nor practical guidelines for preventing and treating DPM.

Specific Aims: The investigators currently are assessing the neural reward system in subjects with perimenopausal major depressive disorder (PM-MDD) and those without depression ("controls") using functional magnetic resonance imaging (fMRI) at baseline and following estrogen replacement therapy (ERT). The Foundation of Hope (FOH) award will allow us to add a Tissue Selective Estrogen Complex (TSEC) treatment condition in a separate group of PM-MDD. The investigators' central hypothesis is that the neural reward system is hypoactive in PM-MDD, and the antidepressant effects of a three-week TSEC intervention will be associated with increased activity in the neural reward system, assessed using functional magnetic resonance imaging (fMRI). The investigators will test the hypothesis by executing the following aims: Aim 1: Determine the extent to which TSEC reduces anhedonia and other depressive symptoms in PM-MDD. Anhedonia and other depressive symptoms will be assessed at baseline and following TSEC administration. The investigators also will compare the effects of TSEC and ERT in PM-MDD. Hypothesis 1: Women PM-MDD will report a significant reduction in depressive symptoms following TSEC administration, and the degree of symptom improvement will be associated with the change in frontostriatal responsivity to reward. Aim 2: Quantify the effect of TSEC on the neural reward system in PM-MDD. The investigators will use fMRI at baseline and following TSEC treatment in PM-MDD to probe frontostriatal reward circuitry. The investigator will also compare the effects of TSEC and ERT in PM-MDD. Hypothesis 2: PM-MDD will show increased activation of the frontostriatal circuit in response to reward following TSEC administration (compared with baseline).

ELIGIBILITY:
Inclusion Criteria:

Perimenopause Status: The investigators will employ the Stages of Reproductive Aging Workshop (STRAW) criteria to confirm perimenopausal status. The stages are primarily based on the characteristics of the menstrual cycle and secondarily on follicle stimulating hormone (FSH) levels. The anchor for the staging system is the last menstrual period (LMP). The investigators will enroll women who have > 2 skipped cycles with an interval of amenorrhea > 60 days and FSH values > 14, consistent with the late menopause transition (stage-1)*. Women who have taken oral contraceptives continuously for relief of perimenopausal symptoms will be exempt from our LMP criteria, and their perimenopausal status will be determined by FSH alone. Because extremes of body weight (BMI < 18 or > 35 kg/m2) or a history of chronic menstrual cycle irregularity can contribute to inaccurate reproductive staging, these will serve as additional exclusion criteria.

MDD Eligibility Criteria: Current diagnosis of MDD with an onset associated with menstrual cycle irregularity. Present or past mania, psychosis, suicide attempts, and alcohol or drug dependence, and current substance abuse, as determined by the Structure Clinical Interview for The Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) for Axis I Disorders (SCID) are exclusionary.

* Per the STRAW criteria, FSH values are highly variable in the late menopausal transition (stage -1), and clinicians should "carefully evaluate the appropriate FSH value, depending on the assay they use" (Harlow et al, 2012). For nearly two years following the LMP, FSH values can fluctuate between levels characteristic of the early reproductive years and levels characteristic of menopause (Hale et al, 2014). McLendon Labs at the University of North Carolina at Chapel Hill (UNC) uses an FSH assay that defines levels consistently above ? 21.5 IU/mL as post-menopausal (McLendon Labs, 2016). As FSH values do not stabilize at consistently high levels until post-menopause, the investigators are setting our minimum required FSH value at > 14 IU/mL to carefully select for women in the perimenopause transition.

Exclusion Criteria:

* Patients will not be permitted to enter this protocol if they have any of the following:

  1. current medication use (i.e., psychotropics, anti-hypertensives, statins, hormonal preparations, or frequent use of anti-inflammatory agents (> 10 times/month)). Women will be allowed to enroll who take medications without known mood effects (e.g. stable thyroid hormone replacement and occasional (< 5 times/month) use of Ambien);

     * all reported prescription medications will be reviewed and cleared by a study physician prior to a participant's enrollment;
  2. pregnant, breastfeeding or trying to conceive;
  3. LMP more than 12 months prior to enrollment;

     * women who have recently taken oral contraceptives continuously for relief of perimenopausal symptoms will be exempt from the final menstrual period (FMP) criteria, and instead, the presence of menstrual irregularity prior to the use of oral contraceptives and elevated FSH will be used to determine their perimenopausal status;
  4. history of undiagnosed vaginal bleeding;
  5. undiagnosed enlargement of the ovaries;
  6. polycystic ovary syndrome;
  7. history of breast or ovarian cancer;
  8. first degree relative with ovarian cancer;
  9. first degree relative with premenopausal onset or bilateral breast cancer;
  10. 2+ first degree relatives with breast cancer (regardless of onset);
  11. 3+ relatives with postmenopausal breast cancer;
  12. abnormal finding in a provider breast exam and/or mammogram;

      * participants will be given the opportunity to describe these conditions in the online screening survey. Reported conditions that were acute in nature and have resolved completely (as indicated by the medical record or follow-up testing) and/or benign will be reviewed by a study physician prior to enrollment. All chronic conditions will be exclusionary.
  13. known carrier of BRCA1 or 2 mutation;
  14. endometriosis;
  15. blood clots in the legs or lungs;
  16. porphyria;
  17. diabetes mellitus;
  18. malignant melanoma;
  19. Hodgkin's disease;
  20. recurrent migraine headaches that are preceded by aura;
  21. gallbladder or pancreatic disease;

      * participants will be given the opportunity to describe these conditions in the online screening survey. Reported conditions that were acute in nature and have resolved completely (as indicated by the medical record or follow-up testing) and/or benign will be reviewed by a study physician prior to enrollment. All chronic conditions will be exclusionary.
  22. heart or kidney disease;

      * participants will be given the opportunity to describe these conditions in the online screening survey. Reported conditions that were acute in nature and have resolved completely (as indicated by the medical record or follow-up testing) and/or benign will be reviewed by a study physician prior to enrollment. All chronic conditions will be exclusionary.
  23. liver disease;
  24. cerebrovascular disease (stroke);
  25. current cigarette smoking;
  26. current suicidal ideation, mania, psychosis, or alcohol/drug abuse/dependence;
  27. past suicide attempts, mania, alcohol/drug dependence, or psychotic episodes;
  28. chronic depression (i.e., episode(s) lasting 3+ years);
  29. depressive episode(s) within 2 years of enrollment;
  30. self-reported claustrophobia;
  31. peanut allergy;
  32. HIV/AIDS

Ages: 44 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men will not be included in this study, given the stated purpose of studying hormone therapy in perimenopausal women.
Enrollment: 20 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal E Schiller, PhD, Principal Investigator — UNC Dept of Psychiatry
Locations (1):
- University of North Carolina at Chapel Hill School of Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] Kessler RC. Epidemiology of women and depression. J Affect Disord. 2003 Mar;74(1):5-13. doi: 10.1016/s0165-0327(02)00426-3. PMID 12646294
- [Background] Schiller CE, Johnson SL, Abate AC, Schmidt PJ, Rubinow DR. Reproductive Steroid Regulation of Mood and Behavior. Compr Physiol. 2016 Jun 13;6(3):1135-60. doi: 10.1002/cphy.c150014. PMID 27347888
- [Background] Schmidt PJ, Haq N, Rubinow DR. A longitudinal evaluation of the relationship between reproductive status and mood in perimenopausal women. Am J Psychiatry. 2004 Dec;161(12):2238-44. doi: 10.1176/appi.ajp.161.12.2238. PMID 15569895
- [Background] Schmidt PJ, Nieman L, Danaceau MA, Tobin MB, Roca CA, Murphy JH, Rubinow DR. Estrogen replacement in perimenopause-related depression: a preliminary report. Am J Obstet Gynecol. 2000 Aug;183(2):414-20. doi: 10.1067/mob.2000.106004. PMID 10942479
- [Background] Schmidt PJ, Ben Dor R, Martinez PE, Guerrieri GM, Harsh VL, Thompson K, Koziol DE, Nieman LK, Rubinow DR. Effects of Estradiol Withdrawal on Mood in Women With Past Perimenopausal Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Jul;72(7):714-26. doi: 10.1001/jamapsychiatry.2015.0111. PMID 26018333
- [Background] Forbes EE, Hariri AR, Martin SL, Silk JS, Moyles DL, Fisher PM, Brown SM, Ryan ND, Birmaher B, Axelson DA, Dahl RE. Altered striatal activation predicting real-world positive affect in adolescent major depressive disorder. Am J Psychiatry. 2009 Jan;166(1):64-73. doi: 10.1176/appi.ajp.2008.07081336. Epub 2008 Dec 1. PMID 19047324
- [Background] Bless EP, McGinnis KA, Mitchell AL, Hartwell A, Mitchell JB. The effects of gonadal steroids on brain stimulation reward in female rats. Behav Brain Res. 1997 Jan;82(2):235-44. doi: 10.1016/s0166-4328(96)00129-5. PMID 9030405
- [Background] Schiller, C. The hormone withdrawal hypothesis of postpartum depression: a translational approach. Theses Diss. (2011).
- [Background] Thomas J, Metereau E, Dechaud H, Pugeat M, Dreher JC. Hormonal treatment increases the response of the reward system at the menopause transition: a counterbalanced randomized placebo-controlled fMRI study. Psychoneuroendocrinology. 2014 Dec;50:167-80. doi: 10.1016/j.psyneuen.2014.08.012. Epub 2014 Sep 1. PMID 25222702
- [Background] Kenna HA, Rasgon NL, Geist C, Small G, Silverman D. Thalamo-Basal Ganglia connectivity in postmenopausal women receiving estrogen therapy. Neurochem Res. 2009 Feb;34(2):234-7. doi: 10.1007/s11064-008-9756-z. Epub 2008 Jun 6. PMID 18535904
- [Background] Schmidt PJ, Nieman LK, Danaceau MA, Adams LF, Rubinow DR. Differential behavioral effects of gonadal steroids in women with and in those without premenstrual syndrome. N Engl J Med. 1998 Jan 22;338(4):209-16. doi: 10.1056/NEJM199801223380401. PMID 9435325
- [Background] Pinkerton JV, Thomas S. Use of SERMs for treatment in postmenopausal women. J Steroid Biochem Mol Biol. 2014 Jul;142:142-54. doi: 10.1016/j.jsbmb.2013.12.011. Epub 2013 Dec 25. PMID 24373794
- [Background] U.S. Census Bureau. Age and Sex Composition: 2010. (2011).
- [Background] Gold EB, Bromberger J, Crawford S, Samuels S, Greendale GA, Harlow SD, Skurnick J. Factors associated with age at natural menopause in a multiethnic sample of midlife women. Am J Epidemiol. 2001 May 1;153(9):865-74. doi: 10.1093/aje/153.9.865. PMID 11323317
- [Background] Cohen LS, Soares CN, Vitonis AF, Otto MW, Harlow BL. Risk for new onset of depression during the menopausal transition: the Harvard study of moods and cycles. Arch Gen Psychiatry. 2006 Apr;63(4):385-90. doi: 10.1001/archpsyc.63.4.385. PMID 16585467
- [Background] Bromberger JT, Matthews KA, Schott LL, Brockwell S, Avis NE, Kravitz HM, Everson-Rose SA, Gold EB, Sowers M, Randolph JF Jr. Depressive symptoms during the menopausal transition: the Study of Women's Health Across the Nation (SWAN). J Affect Disord. 2007 Nov;103(1-3):267-72. doi: 10.1016/j.jad.2007.01.034. Epub 2007 Feb 28. PMID 17331589
- [Background] Wassertheil-Smoller S, Hendrix SL, Limacher M, Heiss G, Kooperberg C, Baird A, Kotchen T, Curb JD, Black H, Rossouw JE, Aragaki A, Safford M, Stein E, Laowattana S, Mysiw WJ; WHI Investigators. Effect of estrogen plus progestin on stroke in postmenopausal women: the Women's Health Initiative: a randomized trial. JAMA. 2003 May 28;289(20):2673-84. doi: 10.1001/jama.289.20.2673. PMID 12771114
- [Background] Thase ME, Entsuah R, Cantillon M, Kornstein SG. Relative antidepressant efficacy of venlafaxine and SSRIs: sex-age interactions. J Womens Health (Larchmt). 2005 Sep;14(7):609-16. doi: 10.1089/jwh.2005.14.609. PMID 16181017
- [Background] Grigoriadis S, Kennedy SH, Bagby RM. A comparison of antidepressant response in younger and older women. J Clin Psychopharmacol. 2003 Aug;23(4):405-7. doi: 10.1097/01.jcp.0000085415.08426.c6. PMID 12920418
- [Background] Masand PS, Gupta S. Long-term side effects of newer-generation antidepressants: SSRIS, venlafaxine, nefazodone, bupropion, and mirtazapine. Ann Clin Psychiatry. 2002 Sep;14(3):175-82. doi: 10.1023/a:1021141404535. PMID 12585567
- [Background] Gyllstrom ME, Schreiner PJ, Harlow BL. Perimenopause and depression: strength of association, causal mechanisms and treatment recommendations. Best Pract Res Clin Obstet Gynaecol. 2007 Apr;21(2):275-92. doi: 10.1016/j.bpobgyn.2006.11.002. Epub 2006 Dec 12. PMID 17166771
- [Background] First, M. B., Spitzer, R. L., Gibbon, M. & Williams, J. B. W. Structured Clinical Interview for DSM-IV-TR Axis I Disorders, Research Version, Non-patient Edition. (SCID-I/NP). (Biometrics Research, New York State Psychiatric Institute, 2002).
- [Background] Harlow SD, Gass M, Hall JE, Lobo R, Maki P, Rebar RW, Sherman S, Sluss PM, de Villiers TJ; STRAW + 10 Collaborative Group. Executive summary of the Stages of Reproductive Aging Workshop + 10: addressing the unfinished agenda of staging reproductive aging. Fertil Steril. 2012 Apr;97(4):843-51. doi: 10.1016/j.fertnstert.2012.01.128. Epub 2012 Feb 16. PMID 22341880
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Watson D, O'Hara MW, Simms LJ, Kotov R, Chmielewski M, McDade-Montez EA, Gamez W, Stuart S. Development and validation of the Inventory of Depression and Anxiety Symptoms (IDAS). Psychol Assess. 2007 Sep;19(3):253-68. doi: 10.1037/1040-3590.19.3.253. PMID 17845118
- [Background] Clark LA, Watson D, Mineka S. Temperament, personality, and the mood and anxiety disorders. J Abnorm Psychol. 1994 Feb;103(1):103-16. PMID 8040472
- [Background] Greene JG. Constructing a standard climacteric scale. Maturitas. 2008 Sep-Oct;61(1-2):78-84. doi: 10.1016/j.maturitas.2008.09.011. PMID 19434881
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Knutson B, Fong GW, Adams CM, Varner JL, Hommer D. Dissociation of reward anticipation and outcome with event-related fMRI. Neuroreport. 2001 Dec 4;12(17):3683-7. doi: 10.1097/00001756-200112040-00016. PMID 11726774
- [Background] Dichter GS, Kozink RV, McClernon FJ, Smoski MJ. Remitted major depression is characterized by reward network hyperactivation during reward anticipation and hypoactivation during reward outcomes. J Affect Disord. 2012 Feb;136(3):1126-34. doi: 10.1016/j.jad.2011.09.048. Epub 2011 Oct 28. PMID 22036801
- [Background] Harlow SD, Gass M, Hall JE, Lobo R, Maki P, Rebar RW, Sherman S, Sluss PM, de Villiers TJ; STRAW 10 Collaborative Group. Executive summary of the Stages of Reproductive Aging Workshop + 10: addressing the unfinished agenda of staging reproductive aging. Menopause. 2012 Apr;19(4):387-95. doi: 10.1097/gme.0b013e31824d8f40. PMID 22343510
- [Background] Hale GE, Robertson DM, Burger HG. The perimenopausal woman: endocrinology and management. J Steroid Biochem Mol Biol. 2014 Jul;142:121-31. doi: 10.1016/j.jsbmb.2013.08.015. Epub 2013 Oct 14. PMID 24134950
- [Background] McLendon Labs. (2016). Follicle Stimulating Hormone (FSH). Retrieved from: http://www.uncmedicalcenter.org/mclendon-clinical-laboratories/available-tests/follicle-stimulating-hormone-fsh/
- [Background] Santen RJ, Allred DC, Ardoin SP, Archer DF, Boyd N, Braunstein GD, Burger HG, Colditz GA, Davis SR, Gambacciani M, Gower BA, Henderson VW, Jarjour WN, Karas RH, Kleerekoper M, Lobo RA, Manson JE, Marsden J, Martin KA, Martin L, Pinkerton JV, Rubinow DR, Teede H, Thiboutot DM, Utian WH; Endocrine Society. Postmenopausal hormone therapy: an Endocrine Society scientific statement. J Clin Endocrinol Metab. 2010 Jul;95(7 Suppl 1):s1-s66. doi: 10.1210/jc.2009-2509. Epub 2010 Jun 21. PMID 20566620
- [Background] ACOG Practice Bulletin No. 141: management of menopausal symptoms. Obstet Gynecol. 2014 Jan;123(1):202-216. doi: 10.1097/01.AOG.0000441353.20693.78. PMID 24463691
- [Derived] Nathan MD, Bondy E, Prim J, Gibson K, Rubinow DR, Meltzer-Brody S, Schiff LD, Carey ET, Schiller CE. Characterizing the spectrum of distress symptoms in midlife women with perimenopausal depression. J Affect Disord. 2026 Jan 1;392:120219. doi: 10.1016/j.jad.2025.120219. Epub 2025 Sep 3. PMID 40912312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process included, social media advertising using Facebook, Instagram, and Craigslist; mass emailing using university wide emails and a database of select University of North Carolina (UNC) healthcare patients (Carolina data warehouse); and flyer advertisements placed in university buildings and local businesses
Pre-assignment Details: Consented participants complete a screening phase that includes a psychiatric interview and gynecological exam prior to the start of study intervention.
Period: Overall Study
Arm/Group | Perimenopausal Women, Depressed
Started | 20
Consented | 20
Received Intervention | 10
Completed | 10
Not Completed | 10
Not completed — Physician Decision | 9
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Perimenopausal Women, Depressed
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 49.9 [44 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian, Non-Hispanic | 15
  Black or African American | 3
  Multi-Racial | 1
  White or Caucasian, Hispanic | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Frontostriatal Reactivity to Reward During MID fMRI Task
Description: The primary outcome measure is functional magnetic resonance imaging (fMRI) data collected during a Monetary Incentive Delay (MID) Task. All participants will complete the fMRI Monetary Incentive Delay (MID) task at baseline and at 3 weeks. During the task, participants need to select the correct response during "win" and "lose" conditions by pressing a button on a button box in the MRI. Participant's blood-oxygen-level dependent (BOLD) activation response (A measurement of oxygen level that is released to neurons since areas of the brain that are thought to be more "active" or involved in certain tasks require more oxygen to perform the tasks.) is measured while they performed the task in MRI scanner.
Time Frame: Baseline to 3 weeks
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Perimenopausal Women, Depressed
Number analyzed (Participants) | 10
percent signal change
  Caudate Baseline | .0704 (.0796)
  Caudate Posttreatment | .0475 (.0692)
  Nucleus Accumbens Baseline | .0623 (.0549)
  Nucleus Accumbens Posttreatment | .0280 (.1166)
  Putamen Baseline | .0399 (.0459)
  Putamen Posttreatment | .0408 (.0823)
Statistical Analysis 1: Comparison: Perimenopausal Women, Depressed; [Ho]: TSEC has no meaningful effect on activity within key nodes of the frontostriate in response to reward; Test type: Non-Inferiority — For analyses the researchers used a paired T-test to compare baseline and post-treatment mean activation values across 3 regions of interest (ROIs): the caudate, putamen and nucleus accumbens; p = 0.53, t-test, 2 sided

2. Primary Outcome: Depressive Symptoms as Measured by the MASQ-AD
Description: The second primary outcome measure uses the Mood and Anxiety Symptoms Questionnaire - Anhedonic Depression Scale (MASQ-AD) to examine symptom change. All participants will complete the MASQ-AD at each study visit, which measures their current symptoms of depression and anxiety. Scores range from 22 to 110 with lower scores reflecting a better outcome.
Time Frame: Baseline, week 2, week 3, week 4 (post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Perimenopausal Women, Depressed
Number analyzed (Participants) | 10
score on a scale
  Baseline Week 1 | 72.1 (9.7)
  Week 2 | 62.4 (13.24)
  Week 3 | 57.2 (11.57)
  Post Treatment Week 4 | 54.5 (10.83)
Statistical Analysis 1: Comparison: Perimenopausal Women, Depressed; [Ho] No change in depressive symptoms from baseline throughout 3 weeks of TSEC administration; Test type: Non-Inferiority — Analysis included MASQ-AD scores from all visits to characterize the change in scores from baseline to post-treatment; p < 0.001, GLM — Mixed models of 3 week TSEC administration for MASQ-AD scores assessed at each study visit from baseline to post-treatment; GLM = -5.8, Standard Error of Mean 1.59 — F value=13.26

ADVERSE EVENTS:
Time Frame: Adverse event data was tracked from the time participants started the intervention through the end of the protocol (approximately 1 month).
Description: All adverse events were tracked by the investigator until the events were resolved, the subject was lost to follow-up, or the adverse event was otherwise explained.
Arm/Group | Perimenopausal Women, Depressed
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perimenopausal Women, Depressed (N=10)
Bloating (Endocrine disorders) | 3 (3)
Hot Flashes (Endocrine disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (4)
Cramps (Reproductive system and breast disorders) | 2 (2)
Heavy Menses (Reproductive system and breast disorders) | 2 (2)
Spotting (Reproductive system and breast disorders) | 2 (2)
Night Sweats (Endocrine disorders) | 1 (1)
Appetite Increase (Endocrine disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Increase in Ear Wax (Ear and labyrinth disorders) | 1 (1)
Toothache (General disorders) | 1 (1)
Poison Ivy Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Numbness and Tingling (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT03740009/Prot_SAP_000.pdf